CLINICAL TRIAL: NCT00341406
Title: Adipose Cell Size In Human Insulin Resistance
Brief Title: Fat Cell Size in Insulin Resistance
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903290; 03-DK-N290
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: Multisizer 3; Signaling; Obesity; Type 2 Diabetes; Adipose Cell Turn Over
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Healthy volunteers: healthy, non-overweight or other medical conditions
- Patients overweight: Those who are generally healthy but overweight
- Patients with health conditions: Those with diabetes and cardiovascular disease.

SUMMARY:
This study, conducted at Stanford University in Palo Alto, California, will examine how insulin metabolism and cardiovascular risk are altered in response to weight loss. Insulin is a natural hormone that causes cells to remove glucose (sugar) from the blood. People who are insulin-sensitive remove glucose efficiently. People who are insulin-resistant require more insulin to remove glucose from the blood.

Adult volunteers will be recruited for this study through advertisements in local newspapers in communities around Stanford University.

Participants will undergo the following tests and procedures:

* Insulin sensitivity testing: Before beginning the study, participants will be tested for insulin sensitivity. For the test, two small catheters (plastic tubes) are placed into two veins - one for infusing glucose, insulin, and sandostatin (a drug that blocks insulin secretion from the pancreas), and one for drawing blood samples. The infusions are done over 3 hours. Blood samples are collected before, during, and at the end of the study to measure how well the cells remove glucose from the blood in response to insulin.
* Research diet: Participants are assigned to a low-calorie diet tailored to the individual's metabolic rate. The diets contain either 40 or 60 percent of total calories as carbohydrates, 40 or 20 percent as fat, and the rest as protein. People with type 2 diabetes who are taking diabetes medicine with have a diet of 45 to 50 percent carbohydrates, 35 to 40 percent fat, and the rest protein.
* Meal profile: Before beginning the diet and after 4 months on the diet, participants are tested for the effects of the various study diets on control of blood sugar and fats. On the day of each test, participants have a physical examination and provide a medical history. Then, a small catheter is placed in a vein. Blood samples are drawn before breakfast and then hourly for up to 8 hours.
* Participants who are diabetic are randomly assigned to take one of three diabetes medications - rosiglitazone, glucophage, or a sulfonylurea compound - to help control blood glucose levels.
* Magnetic resonance imaging: This diagnostic test uses a strong magnetic field and radio waves to show structural and chemical changes in tissues. During the scan, the participant lies on a table in a narrow cylinder containing a magnetic field, wearing ear plugs to muffle loud knocking and thumping sounds that occur during the scanning process. He or she can speak with a staff member via an intercom system at all times during the procedure.

In addition to these procedures, patients may be asked to have a fat cell biopsy. This is done to determine whether insulin-resistant people have fewer fat cells but more fat per cell than insulin-sensitive people. For this test, a small piece of fat tissue is surgically removed, under local anesthetic, from an area of the lower abdomen. With the participant's consent, genetic testing may be done on the fat tissue sample to look for genes that may link central obesity to insulin resistance.

Some participants may be asked to be followed for an additional 3 months after completion of the study for a continued weight loss program. The follow-up includes weekly visits for weight measurements and a review of food records.

DETAILED DESCRIPTION:
Little is known about the turnover of adipose cells in the fat depots of normal animals and human subjects. However, microarray analysis of adipose cell gene expression in high risk insulin-resistant human subjects suggests that a reduced rate of adipose cell turnover is associated with enhanced adipose cell size and systemic insulin resistance. New technology now permits a detailed analysis of adipose cell size including the detection of smaller cells which may be in the process of active differentiation. We propose to examine the relationship between adipose cell size distribution and systemic insulin resistance in obese human subjects. Adipose tissue biopsies will be obtained at Stanford University under protocols and consent forms approved by the Stanford University IRB. Only procedures already being performed on subjects under these protocols will be used.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Without regard to gender, race, or socioeconomic status, all subjects will be adult men and women. The racial/ethnic composition of the study population will be reflective of the communities surrounding Stanford University. Subjects will be recruited through placement of advertisements in local newspapers, but no subjects will be seen at NIH.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The NIH is involved with several Stanford protocols that have recruited both males & females between ages of 40-65 years of age who are either overweight patients but generally healthy, those with diabetes and cardiovascular medical conditions and/or are healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 782 (Actual)
Dates: Start 2003-09-04 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
adipose cell size distribution | end of study
  to look at role of the to look at role of the fat cell in relation to obesity and insulin resistance, the role of anti-inflammatory helper cells in protecting against insulin resistance, look at effects of overfeeding on fat cells and insulin resistance, measure inflammatory markers (during and after weight loss), quantify production of fat cells, total triglycerides production, and breakdown of fat cells.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Sherman, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Disorders (NIDDK), 9000, Bethesda, Maryland, United States